CLINICAL TRIAL: NCT00550186
Title: The Effect of Intravascular Preload on Bladder Retention Volume During Spinal Anesthesia Induced Detrusor Blockade
Brief Title: Effect of Preload on Bladder Retention Volume During Spinal Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rijnstate Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: LTC-420-071206
Record Dates: First submitted 2007-10-26; First posted 2007-10-29 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: Diuresis; Bladder Retention Volume; Hypotension
Keywords: spinal anesthesia; preload; diuresis; bladder retention
MeSH Terms: conditions — Hypotension; Urinary Retention | interventions — Ringer's Lactate

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Placebo Comparator): No preload
  Interventions: Other: placebo
- 2 (Active Comparator): Preload with cristalloid infusion
  Interventions: Drug: Ringers Lactate
- 3 (Active Comparator): Preload with collid infusion
  Interventions: Drug: HaemoHES 6%

INTERVENTIONS:
Other: placebo
  Arms: 1
Drug: Ringers Lactate
  Arms: 2
Drug: HaemoHES 6%
  Arms: 3

SUMMARY:
The purpose of this study is to assess the influence of different fluid infusions on the quantity of bladder retention after spinal anesthesia. This study should determine if this increase in bladder retention is significant and relevant.

DETAILED DESCRIPTION:
Background of the study:

Spinal anesthesia , through interruption of spinal nerve conduction, causes intense blockade of sensation, motor function as well as (para)sympathetic function. Loss of sympathetic tone causes vasodilation which may lead to arterial hypotension and bradycardia. To avoid these effects, in anesthetic practice, usually intravenouspreload is administered as cristalloids or colloids. The form and dosage of these plasma expanders will influence diuresis during spinal anesthesia-induced detrusor blockade. Excess diuresis may cause bladder distension and neccecitates bladder catheterization

Objective of the study:

To compare the quantitative effects of Ringer Lactate and HES 6% on diuresis during spinal anesthesia-induced detrusor blockade as well as prevention of hypotension and vasopressor use.

Study design:

Before spinal anesthesia is performed, patients are randomized into one of the 3 study groups (no preload, preload with Ringers' Lactate 14 ml/kg, preload with HES 6% 7 ml/kg). Spinal anesthesia is administerd with lidocaine 2% 70mg. Hypotension is treated with vasopressors, atropine or additional intravenous fluid. Bladder scans will be performed on the recovery unit and day-case unit. Total urinary volume is measured until sensory function at dermatome S2/3 is restored and spontanous voiding is possible.

Study population:

ASA 1-2 patients who present for spinal anesthesia for minor surgery on the lower extremitiy. Age 18-60 years.

Intervention (if applicable):

Prespinal administration of intravenous Ringers' Lactate 14 ml/kg or HES 6% 7 ml/kg.

Primary study parameters/outcome of the study:

Primary outcome is total urinary volume during spinal induced detrusor blockade, and number of subjects that have a bladdder volume over 500ml.

Secundary study parameters/outcome of the study (if applicable):

Secondary outcome parameters:

Periods of hypertension, and total dose of vasopressor en extra fluid administration.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness (if applicable):

Except for extra bladderscan and block height measurements, all actions are part of routine anesthesiologic care.

Ga naar boven

ELIGIBILITY:
Inclusion Criteria:

* ASA1-2
* undergoing minor procedure under spinal anesthesia

Exclusion Criteria:

* ASA3-4
* History or signs of heart failure / coronary artery disease.
* Bladder / urinary disease
* Neurologic disease that may affect bladder function

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 144 (Actual)
Dates: Start 2007-10; Primary Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marco Peters, MD, Principal Investigator — Nijmegen University Anesthesiology Department (resident); Ed Kamphuis, Md, PhD, Principal Investigator — Rijnstate Hospital
Locations (1):
- Ziekenhuis Zevenaar, Zevenaar, Gelderland, Netherlands